CLINICAL TRIAL: NCT04436939
Title: Soft Tissue Response to Polyetheretherketone (PEEK) and Titanium (Ti) Healing Abutments on Dental Implants
Brief Title: Soft Tissue Response to Peek and Ti Healing Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Iva Milinkovic, Assistant Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22101980.1
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Dental Implants
Keywords: dental implant; healing abutment; PEEK; Titanium
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: This was a split mouth study design in which both test and control group were the same patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK healing abutment (Experimental): Healing abutment made of polyetheretherketone (PEEK)
  Interventions: Device: Dental implant
- Ti healing abutment (Active Comparator): Healing abutment made of titanium (Ti)
  Interventions: Device: Dental implant

INTERVENTIONS:
Device: Dental implant — Following dental implant installation, PEEK or Ti healing abutments were placed according to the split mouth study design.

SUMMARY:
Introduction: Single-stage dental implant placement protocol involves the placement of healing abutments. In addition to osseointegration process, healing of peri-implant soft tissues is of a great importance too. Routinely, healing abutments made of titanium (Ti) are used. The aim is to find novel materials that would have the same mechanical properties, but less prone to plaque-adhesion and therefore showing lower local inflammatory soft tissue response. Polyetheretherketone (PEEK) is a thermoplastic polymer that has favorable mechanical characteristics, high biocompatibility and low submissiveness to microorganism adhesion. White color makes it aesthetically acceptable in the treatment of patients with thin gingival phenotype.

The Aim: To compare the formation of dental plaque on PEEK and Ti healing abutments and examine the local response of peri-implant tissues.

Materials and Methods: The study included 11 patients with at least two missing teeth in the posterior regions. In each patient, 2 implants were installed, with PEEK abutment (experimental group) placed on one implant, while on the other implant, Ti abutment (control group) was placed. Before prosthetic rehabilitation of patients, both abutments were replaced with new ones and a thin layer of peri-implant soft tissue was sent to histological analysis.

Results: The average age of patients was 49 years. Out of 11 patients, 27% were female and 73% male. 36% of respondents were smokers. Histological immunohistochemical analysis of samples of peri-implant soft tissues showed massive inflammatory infiltration in subepithelial tissue in the experimental group (10/11), while the inflammatory infiltrate in the control group was classified as moderate (7/11) or weak (4/11).

Conclusion: Both types of healing abutments have been shown to be successful in single-stage implantation protocol. However, contrary to expectations and preliminary findings from the literature, PEEK healing abutments showed a more pronounced inflammatory response of the surrounding soft tissues relative to Titanium abutments.

DETAILED DESCRIPTION:
Study design This study was performed at Department of Periodontology and Oral medicine of the Belgrade School of Dental Medicine in collaboration with the Institute of Pathology of the Belgrade School of Medicine. The study was approved by the Institutional Ethical Committee and all subjects enrolled in this trial have signed an informed consent according to the Helsinki declaration of 1964 and subsequent amendments. It was a randomized clinical trial, with a split mouth design, in which each subject served as both experimental and control group.

Study sample The subjects included in this study are patients of the Department of Periodontology and Oral Medicine, School of Dental Medicine, University of Belgrade. Individuals diagnosed with partial edentulism in posterior maxillary or mandibular arches, with missing at least two teeth that were extracted at least 6 months earlier, have been selected following clinical and radiological examination.

Ten patients with indication for implant placement (presenting bilateral single tooth gaps and/or extended edentulous spaces distally from maxillary or mandibular canines) were included in this study if they fulfilled the following criteria:

1. Men and non-pregnant women, 18 to 70 years of age;
2. Systemically healthy patients
3. Adequate bone quantity at the experimental sites to allow the insertion of 3.8 or 4.3 mm diameter implants
4. Sufficient band of keratinized mucosa at the experimental sites
5. No active periodontal disease at the time of inclusion/surgery and proper oral hygiene defined by bleeding on probing scores (BOP) and plaque indices (PI) less then 15%

Titanium implants placed in the posterior mandible and maxilla were randomly assigned to receive transmucosal healing by either: PEEK healing abutment (A, experimental group) or Ti healing abutment (B, control group). Randomization was performed by a toss of a coin.

Surgical procedures

Implant placement was carried out under local anesthesia (2% lidocaine with epinephrine, 1:100000). Mid-crestal incisions were made and mucoperiosteal flaps (MPFs) were elevated not to interfere with muco-gingival junction. Surgical implant sites were prepared according to a standard procedure using a low-trauma surgical technique under copious irrigation with sterile 0.9% physiological saline. Thereafter, two bone level implants were inserted (C-TECH Esthetic line (EL), Italy) in 1mm subcrestally, in a one-stage protocol. The diameter and length of the implant were chosen following CBCT data analysis. Study abutments (C-TECH, Italy) were provided in width of 4 mm and in different heights (2, 3, 4 mm). In the experimental group, immediately following implant placement, a PEEK abutment was screwed at 10 Ncm, while in the control group, the same procedure was performed by means of TI healing abutment.

All abutments were connected using a torque of 10 Ncm. Subsequently, the MPFs were repositioned and adapted using non-resorbable single sutures to ensure a transmucosal healing procedure.

Postoperative Care

Patients were prescribed antimicrobials (Amoxicillin caps. 500mg, 3x1 or Clindamycin, 600mg, 2x1, for patients allergic to penicillin), analgesics (Ibuprofen, 600 mg, every 6 hours) and 0.2% chlorhexidine solution (ASD Curasept 212, Curaden, Switzerland). Sutures were removed one week after the surgery.

Sampling 3 months following the implant surgery, a minimally invasive surgical procedure was performed for the placement of larger diameter (5mm wide) healing abutments. At this stage, a triangular incision was performed at mesial and distal aspect of the existing implant healing abutment, to remove both the healing abutment with the band of the surrounding soft tissue of 1-1.5mm in thickness.

Soft tissue specimens were gently rinsed with 4% formalin and fixed in 4% neutral buffered formalin solution. The samples were processed to the laboratory for further histological preparation.

Finally, commercially available 5 mm wide healing abutments (C-TECH) were selected by height according to the individual situation and applied to ensure a conditioning of the soft tissues prior to prosthetic restauration.

Light microscopic analysis Analysis was performed by two independent observer-pathologists, blinded to the treatment, samples marked as patients from group A and B. For microscopic histological evaluation, biopsy were fixed in 10% neutral-buffered formalin. Three 5-μm-thick paraffin-embedded horizontal sections were cut dyed with a haematoxylin-eosin (HE) stain and analyzed by light microscopy and microscope Nikon Eclipse Ci with control unit DS-L3 and pre-installed software. Following morphological changes were analyzed: presence, localization and intensity of the inflammation. Presence in epithelial and subepithelial tissue were categorized qualitatively (yes/no) and intensity semiqualitatively (light, medium, intensive).

For immunohistochemical analysis serial sections, 5 µm thick, were cut and immunohistochemical techniques were carried out using the avidin-biotin-peroxidase complex method with an LSAB2 kit (Dako, Glostrup, Denmark). The primary antibodies used in this study were: LCA (M3629Clone 318-6-11, dilution 1 : 25; Dako), CD 3 (M3539 Clone β-catenin1, dilution 1 : 200; Dako), CD 20 (M7240 Clone MIB-1, dilution 1 : 100; Dako), and CD 68 (EPR2241, ab134175, dilution 1 : 200; Abcam).

Cells with cytoplasmic staining were considered positive in immunohistochemistry for all antibodies. The labeled-cell count of all antibodies was determined in ten high-power fields at 200× magnification.

In statistics, uni- and multivariate analyses were used, and a p-value of less than 0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with partial edentulism in posterior maxillary or mandibular arches, with missing at least two teeth that were extracted at least 6 months earlier
* Adequate bone quantity at the experimental sites to allow the insertion of 3.8 or 4.3 mm diameter implants
* Sufficient band of keratinized mucosa at the experimental sites
* No active periodontal disease at the time of inclusion/surgery and proper oral hygiene defined by bleeding on probing scores (BOP) and plaque indices (PI) less then 15%

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Soft tissue inflammatory reaction around healing abutments | Three month after the implant placement
  For microscopic histological evaluation, soft tissue biopsies were prepared, dyed with a haematoxylin-eosin stain and analyzed by light microscopy for presence, localization and intensity of the inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Zoran M Aleksic, DDS, MS, PhD, Study Director — Department of Periodontology, Belgrade School of Dental Medicine
Locations (1):
- Department of Periodontology, School of Dental Medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milinkovic I, Krasavcevic AD, Jankovic S, Sopta J, Aleksic Z. Immunohistochemical analysis of soft tissue response to polyetheretherketone (PEEK) and titanium healing abutments on dental implants: a randomized pilot clinical study. BMC Oral Health. 2022 Nov 11;22(1):484. doi: 10.1186/s12903-022-02536-0. PMID 36368972